CLINICAL TRIAL: NCT04574856
Title: A Phase II Study of Multiparametric MR-Guided High Dose Adaptive Radiotherapy With Concurrent Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Multiparametric MR-Guided High Dose Adaptive Radiotherapy With Concurrent Temozolomide in Patients With Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2020.033; HUM00179427 (Other: University of Michigan)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Patients with Newly Diagnosed Glioblastoma (Experimental): Patients will receive dose-intensified, adaptive photon radiation therapy
  Interventions: Radiation: Dose-Intensified Radiotherapy; Drug: Temozolomide; Drug: Adjuvant temozolomide

INTERVENTIONS:
Radiation: Dose-Intensified Radiotherapy — Adaptive, dose-intensified radiotherapy targeting an advanced imaging signature, with a target, nominal radiotherapy dose of 80 Gy.
Drug: Temozolomide — Temozolomide chemotherapy (75 mg/m2 daily for 6 weeks)
Drug: Adjuvant temozolomide — Adjuvant temozolomide will be delivered at 150-200 mg/m2 days 1-5 every 28 days for 6 cycles, with additional cycles delivered at the discretion of the investigator.

SUMMARY:
This study will investigate whether or not intensified radiation therapy adapted during the radiation treatment course to high-risk, treatment-resistant tumor regions will improve overall survival in patients with newly diagnosed glioblastoma (GBM) compared to conventional chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Newly diagnosed, histologically-confirmed supratentorial WHO grade IV gliomas including glioblastoma (all variants) and gliosarcoma. Prior low-grade glioma without prior RT, now with malignant progression are eligible.
* Karnofsky performance status >=70
* Minimal life expectancy of 12 weeks
* Adequate bone marrow reserve (Hemoglobin ≥ 10 g/dL, absolute neutrophils ≥ 1500/mm3, platelet count ≥ 100,000/mm3), acceptable liver function (total bilirubin ≤ 2 x upper limit of normal (ULN) (unless elevated bilirubin is related to Gilbert syndrome), and ALT/AST ≤ 5 x ULN) and renal function (serum creatinine ≤ 2.0 mg/dL) within 14 day prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
* Maximal contiguous diameter of tumor based on high b-value diffusion MRI and DCE perfusion MRI ≤5 cm
* Patients must be registered within 6 weeks of most recent resection
* Females of child-bearing potential must have a negative pregnancy test within 14 days prior to registration. Patients with reproductive potential must agree to use an effective contraceptive method during treatment and study participation.

Exclusion Criteria:

* Recurrent glioma, or tumor involving the brainstem or cerebellum
* Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment is not permitted. Prior chemotherapy for a different cancer is allowable if interval since last treatment cycle completion is >3 years.
* Evidence of CSF dissemination (positive CSF cytology for malignancy or MRI findings consistent with CSF dissemination)
* Evidence of severe concurrent disease requiring treatment
* Prior invasive malignancy (except non-melanoma skin cancer or non-life limiting invasive malignancy that may not require treatment, such as low-risk prostate cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of breast, oral cavity or cervix are all permissible)
* Patients unable to undergo MRI exams (i.e. patients with non-compatible devices such as cardiac pacemakers, other implanted electronic devices, metallic prostheses, or ferromagnetic prostheses [e.g. pins in artificial joints and surgical pins/clips], or unable to receive gadolinium for MRI, as per the standard Department of Radiology MRI screening criteria)
* Patients treated with previous cranial or head/neck radiotherapy leading to significant radiation field overlap as determined by treating physician
* Multifocal disease (>1 lobe of involvement) of discontiguous contrast enhancing disease as seen on conventional MRI
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
12-month overall survival rate | 12 months post radiation therapy (RT)
  12-month overall survival rate of study participants (failure defined as death due to any cause)

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival (failure defined as death due to any cause)
Progression-free survival rate | 2 years
  Progression-free survival (failure defined as progression or death due to any cause) will be evaluated using standard response assessment in neuro-oncology (RANO) criteria.
Proportion of failures classified by relation to the high-dose radiation region | 2 years
  Patterns of failure (tumor growth) will be classified as follows:
  * Central: >95% of the tumor volume is within the high-dose radiation region
  * In-field: >80% to 95% of the tumor volume is within the high-dose radiation region
  * Marginal: 20-80% of the tumor volume is within the high-dose radiation region
  * Distant: <20% of the tumor volume is within the high-dose radiation region
Advanced MRI Gross tumor volume (GTV) and its association with overall survival | 3 months post-RT
  GTV is defined as the combined hypercellularity tumor volume and hyperperfused tumor volume, assessed by high b-value diffusion MRI and dynamic contrast-enhanced perfusion MRI, respectively. Patients will be grouped into those with less than 2.5 cc GTV and those with 2.5 cc or more GTV. This measure will be used to determine whether advanced MRI metrics can be used to distinguish pseudoprogression from true tumor progression, and to determine whether advanced MR-identified tumor volume 3 months post-chemoradiation is associated with survival.
Patient-reported quality of life (QOL) using EORTC QLQ-C30 and BN20 | Up to 12 months post-RT
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) is a validated questionnaire developed to assess the quality of life of cancer patients, with the EORTC QLQ-BN20 specifically for brain tumor patients. Patients will be classified as having deterioration if there is a clinically meaningful change (10 point drop from baseline) in the QOL scales. The percentage of patients with deterioration in each survey will be reported.
Patient-reported symptom burden using MDASI-BT | Up to 12 months post-RT
  The MD Anderson Symptom Inventory for Brain Tumor (MDASI-BT) is a validated questionnaire developed to assess the symptom burden of brain tumor patients. Severity of symptoms is scored on a scale of 0-10, with 0 being "not present" and 10 being "as bad as you can imagine." Patients will be classified as having deterioration if there is a clinically meaningful change (1 point increase in symptom severity from baseline). The percentage of patients with deterioration will be reported.
Patient objective neurocognitive function | Up to 12 months post-RT
  Objective neurocognitive function (NCF) testing using Hopkins Verbal Learning Tests, Controlled Oral Word Association, and Trail Making Tests A and B. Test results will be reported as a composite, using the reliable change index (RCI) to categorize patients as improved, stable, or declined from baseline.
Grade 3 or higher treatment-related toxicities | 12 months post-RT
  Rate of grade 3 or higher toxicities (neurologic and non-neurologic) of dose-intensified, adaptive chemoradiotherapy. Toxicity assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kim, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim MM, Aryal MP, Suresh K, Rosen BS, Parmar H, You D, Leung D, Clarke N, Fortunato J, Al-Holou W, Heth J, Altshuler D, Hollon T, Edwards DM, Wahl DR, Lawrence TS, Cao Y. A Phase 2 Study of Multiparametric Magnetic Resonance Imaging-Guided High-Dose Response-Adaptive Radiation Therapy With Concurrent Temozolomide in Patients With Newly Diagnosed Glioblastoma: Results From an Interim Analysis. Int J Radiat Oncol Biol Phys. 2025 Jul 1;122(3):605-610. doi: 10.1016/j.ijrobp.2025.02.020. Epub 2025 Mar 8. PMID 40058709